CLINICAL TRIAL: NCT02476383
Title: Spinal Manipulative Therapy Treatment Effect Modifiers in Individuals With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201400928
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- augmented spinal manipulative therapy (Active Comparator): Participants in this group will receive spinal manipulative therapy provided by a practitioner interacting in a warm and friendly way who is free to respond to participant conversation. Participants in this group will receive information about the effectiveness of spinal manipulative therapy for some individuals experiencing low back pain.
  Interventions: Procedure: spinal manipulative therapy
- neutral spinal manipulative therapy (Active Comparator): Participants in this group will receive spinal manipulative therapy provided by a practitioner engaging in minimal interaction. Participants in this group will not receive information about the effectiveness of spinal manipulative therapy for some individuals experiencing low back pain.
  Interventions: Procedure: spinal manipulative therapy

INTERVENTIONS:
Procedure: spinal manipulative therapy — refer to arm descriptions

SUMMARY:
This study considers whether treatment effects in response to spinal manipulative therapy for individuals experiencing low back pain are dependent upon the context in which the intervention is provided. Half of the participants will receive spinal manipulative therapy with encouragement to interact with the provider and information to enhance expectations for the effectiveness of the intervention. The other half will receive spinal manipulative therapy with minimal interaction with the provider.

ELIGIBILITY:
Inclusion Criteria:

* Currently experiencing low back pain defined as pain located below the 12th rib and above the inferior gluteal fold with or without corresponding leg pain;
* Low back pain symptom intensity rated as 4/10 or higher during the last 24 hour;
* Appropriate for conservative treatment for low back pain.

Exclusion Criteria:

* Non-English speaking;
* Systemic medical conditions know to affect sensation (e.g. diabetes);
* History of lumbar surgery or fracture within the past 6 months;
* Received spinal manipulative therapy for treatment of low back pain within past 6 months;
* Current or history of chronic pain condition other than low back pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
numeric pain rating scale | Change in baseline at 2 weeks
  0 to 100 with 0= no pain at all to 100= worst pain imaginable

SECONDARY OUTCOMES:
Oswestry Disability Index | Change in baseline at 2 weeks
  0 to 100 with 0= no perceived disability to 100= greatest perceived disability
Back Performance Scale | Change in baseline immediately following spinal manipulative therapy during day 1 and at 2 weeks
  0 to 15 with lower scores indicating better performance
Quantitative Sensory Testing | change in baseline immediately following spinal manipulative therapy during day 1
  standardized thermal and pressure stimuli will be applied and participant will rate the pain associated with each using a 0= no pain to 100= worst pain imaginable numeric pain rating scale or a mechanical visual analog scale anchored with no pain and worst pain imaginable
Patient Centered Outcome Questionnaire | change in baseline immediately following spinal manipulative therapy during day 1
  Participants indicate their usual level, desired level, successful level, and expected level of pain, fatigue, emotional distress, and interference using a 0= none at all to 100= worst imaginable numeric rating scale
Working alliance subscale of the Pain Rehabilitation Expectation Scale | change in baseline immediately following spinal manipulative therapy during day 1
  Scored from 16= lesser therapeutic alliance to 64= greater therapeutic alliance
North American Spine Society Lumbar Spine Outcome Assessment | 2 weeks
  Participants will answer 3 questions: 1) If you had to spend the rest of your life with the low back pain you have right now, how would you feel about it? Scored from 1= very dissatisfied to 5= very satisfied; 2) Would you have the same intervention you received in this study again for low back pain? Scored from 1=Definitely not to 5= definitely yes; 3) . How would you rate the overall results of the intervention you received in this study for low back pain? Scored from 1= Terrible to 6= Excellent
Semi- structured qualitative interview seeking insight into answers on the working alliance subscale of the pain rehabilitation expectation scale | 2 weeks
  a brief semi- structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Joel E Bialosky, PT, PhD., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No